CLINICAL TRIAL: NCT06786429
Title: Managing Hepatitis B (Hep. B) and Human Papilloma Virus (HPV) Related Cancers Among Women of Childbearing Age, and Young Adults in Zimbabwe in the Context of Mental Health: a Multimodal, Multifaceted Approach.
Brief Title: Managing Hepatitis B (Hep. B) and Human Papilloma Virus (HPV) Related Cancers and Mental Health.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Dube (Other)
Collaborators: National University of Science and Technology, Zimbabwe (Other)
Responsible Party: Principal Investigator, Eunice Dube, Project Director/Principal Investigator, Eunice Dube
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EX8KG3L2Z649
Record Dates: First submitted 2025-01-13; First posted 2025-01-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B; Human Papilloma Virus; Gall Stones (& [Calculus - Gall Bladder]); Mental Health Issue; Cancer Liver; Cancer of Cervix; Depression, Anxiety
MeSH Terms: conditions — Hepatitis B; Gallstones; Carcinoma, Hepatocellular; Uterine Cervical Neoplasms; Depression; Anxiety Disorders | interventions — Hepatitis B Vaccines; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: High school kids and women of child bearing age are participating concurrently as separate groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High School Students (Other): All high school students in study area are eligible, approximately 1000-1500 students.
  Participants will complete a Youth Risk Behavior Screen (CDC), offer Cognitive Behavioral Therapy if indicated. Participants will be offered a 3-dose series of Gadarsil to protect against HPV.
  Interventions: Biological: Gardasil 9 vaccine; Behavioral: Cognitive Behavioral Therapy
- Women of childbearing age and young adults (Other): This group is at highest risk for having exposure to cervical and liver cancer, gall bladder issues, depression and anxiety. Participants are unlikely to have had vaccines of interest, Hep B. and HPV as status is unknown due to lack of screening and vaccination. Participants in this group with depressive/anxiety symptoms are likely to benefit from CBT intervention
  Interventions: Biological: Gardasil 9 vaccine; Biological: Hepatitis B Virus Vaccine(HBV); Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Biological: Gardasil 9 vaccine — Participants with a valid consent will be offered a three-dose Gardasil 9 series if eligible.
Biological: Hepatitis B Virus Vaccine(HBV) — Participants who do not demonstrate immunity to Hep B antibody marker in their blood, HBsAb and not HBsAg will be offered a three-dose series of Hep B. vaccine. A blood test will be done six months later to assess vaccine take i.e. immunity. Patients who demonstrate infection with Hep B virus will be referred to their doctor for further management.
  Arms: Women of childbearing age and young adults
Behavioral: Cognitive Behavioral Therapy — Participants who demonstrate signs and symptoms of depression and/or anxiety will be offered individual behavioral management services. This consists of weekly individual sessions by a trained therapist for 8 weeks with option for referral for further management depending on the outcome of the intervention. The positive outcome consists of a change in presenting symptoms determined after administration of the youth risk behavior screen for high school students, and PHQ-9, and Edinburgh post-natal depression screen for women respectively.

SUMMARY:
Aim: The main goal of this observational study is to determine the prevalence of Human Papilloma Virus(HPV) infection, and Hepatitis B (Hep B) immunity amongst women of childbearing age 13 to 45 years) attending clinics at Mtshabezi Mission and Matobo clinic respectively; and assess behavioral risk factors of high school students at these catchment areas that can put them at risk for developing cancer of the cervix and liver.

Question: Can screening for cancer, and vaccination against Hep B and HPV, and cognitive behavior intervention help in preventing related cancers amongst these groups of participants.

DETAILED DESCRIPTION:
Hypotheses:

* The prevalence of HPV infection (might be high) and Hep B immunity (might be low) is not documented and therefore unknown in this community as there is no routine surveillance of these specific conditions
* Behavioral risk factors of High School students in Matabeleland South Province have not yet been assessed and remain unaddressed hence the high rates of suicide, infection and teen pregnancy which predispose participants to Hep B and HPV related infection and consequently, cancers. Participants have not had access to the HPV preventing vaccine Gardasil 9. To provide answers to these concerns, investigators propose the activity described below.

Objectives

The objectives of this proposal are twofold:

1. Research- uses the Theory of change and the quantitative epidemiologic descriptive survey method to gather, analyze and interpret data and disseminate results. There is no sampling frame as this study is exploratory. True prevalences are not known.

1.1 Data collection, analysis, and interpretation to determine the burden of HPV infection; determine the HPV types that are prevalent in this community to assess the potential effectiveness of the available vaccine; assess potential for developing vaccine covering local Geno-types, determine the prevalence of immunity to Hep B, assess biliary tract involvement, and depression prevalence among adult participants.1.2 Conduct a youth risk behavior screen to determine potential infection risk and mental health issues, and design intervention strategies.1.3 Disseminate preliminary findings after the first 6 months or year one and suggest intervention strategies that can be evaluated for effectiveness during the study period. Publish findings and scale project to other areas in Zimbabwe and internationally.1.4 Request collaboration with NIH/NCI/Global center/Behavioral health to strengthen research capabilities and service provision in this area.2. Intervention 2.1 Recruit 800 consenting female participants attending prenatal, family planning, post-partum, and other clinics at these selected centers to perform a one-time comprehensive medical exam, pap smear (to detect abnormal cells, and HPV test (if eligible) to detect infection in the cervix); perform blood test to look for Hep. B. and cancer biomarkers' presence, perform a onetime fibro scan and abdominal ultrasound to assess the liver and gall bladder involvement.2.2 Administer the Youth Risk Behavior Screen (Centers for Disease Control and Prevention (CDC) to participating students in the selected schools over a period of 5years to determine the types and significance of problem behavior and suggest appropriate interventions; Assess protective factors among boarders versus day scholars. offer Gardasil 9 vaccine to 1500 eligible students with parental consent over a period of 5 years or until it has been made universally accessible to these participants during the project duration. 2.3 Refer participants with positive screens for further assessments and management including behavioral health intervention as indicated. Assess potential for home visits, telehealth services, routine screening, and immunization to ease access to services. Create teen clinics at the school sites. Analyze data at three levels using the IBM Statistical Package for Social Sciences (SPSS) for significance testing and disseminate results. Solicit Ministry of Health and Childcare (MOHCC) buy-in for scaling to other Provinces.

* Investigators plan to follow-up this cohort, funds permitting, to determine the prevalence of infection with HPV and /or subsequent development of cervical cancer ten years post vaccination with Gardasil 9 vaccine, and 6months to 1 year post Hep B vaccine to determine immunity or infection.
* Based on the data obtained, clinical trials will assess the probability of developing an HPV vaccine that is user and patient friendly to Low to Middle Income Countries (LMIC) countries; promote creation and use of screening tools suitable for rural communities.
* School Behavioral Health services are non-existent currently. It is planned that the introduction of school-based counseling and individualized access to Psychiatric nurse/Psychiatrist/Psychologist will help students stay away from identified risk behaviors that expose them to HPV and other sexually transmitted diseases (STDs), and that HPV vaccine will soon be made universally accessible with help from Global Vaccine Institute (GAVI) and the United States Agency for International Development (USAID).
* Participants identified as having risk behaviors will be offered further assessment by a psychiatrist or /and psychologist to develop a viable framework to prevent and manage such behaviors including medication which is currently not available in Zimbabwe.

Recommendations regarding women's health i.e., screening for cervical cancer and vaccination against HPV and Hep B, depression, Intimate Partner Violence will be guided by the findings of this study.

ELIGIBILITY:
Inclusion Criteria:

* For the High school students' group:

All students aged 13 years and older, enrolled at the selected Mtshabezi and Matopo High Schools in the Gwanda and Matobo Rural Districts during the five-year period of the project are eligible to participate in the study.

Ability to understand and respond to questions on the Youth Risk Behavior Scree questionnaire and PHQ-9 scale.

Relevant history of HPV vaccine administration. Ability to obtain parental/guardian consent for participation.

- For the women group: All women and young female adults thirteen to forty-five years old and requesting health services for prenatal, post-partum, family planning and other care during the five-year project period are eligible to participate.

Must not have received Hep B and HPV vaccine in the past and have no known contraindications to either of these two vaccines.

Are able to understand and respond to the PHQ-9 and Edinburgh Postnatal Depression scales.

Must have a valid consent for participation in the study.

Exclusion Criteria:

* males who are not enrolled in these participating High Schools.
* children below the age of thirteen who are not enrolled in high schools and are not seeking prenatal, post-partum and family planning services at these selected health facilities during the project period.
* Any eligible potential participant without a valid consent.
* Any potential participant who is excluded by a doctor or midwife for a known contraindicating medical condition that can lead to potential harm to the participant or staff.

Any potential participant who is unable to understand and respond to the questions being asked.

Participants with proof of prior vaccination will be excluded from this part of the study.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Human Papilloma Virus infection | Baseline and 10 years post vaccination
  Women will be screened for HPV infection at baseline, and post vaccine with Gardasil 9
Hepatitis B immunity | Baseline and six months to one year post vaccination.
  Women will be screened for Hep B immunity before and after receiving a three-shot series of Hep B vaccine.
cancer of cervix | Baseline assessment and 10 years post vaccination with Gardasil 9.
  Patients will be assessed for malignancy on cervix
Cancer of the liver | Baseline and six months to one year post vaccination with Hep B.
  Patients will have a fibro scan to assess condition of liver at initial visit and post vaccination with Hep B.

OTHER OUTCOMES:
Number of women with gall stones expressed as a rate of total number women examined. | One time at baseline.
  Women will be assessed for gallstones at the initial visit. They will have a onetime abdominal ultrasound to assess the condition of their gall bladder, an important component of the digestive system with close proximity to the liver. Labs reviewed. Poor nutrition is listed among the top ten behavior related causes of mortality in Zimbabwe. There does not appear to be any studies related to the prevalence of this problem in this community. Those with a positive screen will be referred for further management.
A change in Depression and anxiety symptoms based on PHQ-9 and Edinburgh post-natal depression scale. | Baseline and two to 12 months
  Patients undergoing Cognitive Behavioral Therapy will be assessed for change in symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Elopy Sibanda, M.D, Study Director — National University of Science and Technology, Zimbabwe; Eunice Dube, DSc, Principal Investigator — Eunice Dube; Jill Koshiol, Ph. D, Principal Investigator — National Cancer Institute (NCI); Sodumisa Ngwenya, MD, Principal Investigator — Mtshabezi Mission Hospital; Desmond M Kaplan, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
Only test results data with no participant identifying information will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: All selected study supporting information will be available from 01/30/2031 through 01/30/2032.
Access Criteria: Selected IPD will be accessible to researchers at institutes of higher education, NIH, and non-profit organizations through the Zimbabwe data repository.
URL: https://www.nust.ac.zw

REFERENCES:
- See also: tba — https://www.nust.ac.zw
- Available data/document: Clinical Study Report — https://www.nust.ac.zw
- Available data/document: Clinical Study Report: tba — https://www.nust.ac.zw